CLINICAL TRIAL: NCT00830102
Title: A Randomized, Placebo-controlled, Double-blind, Six-way Crossover, Single-dose Exposure Study to Compare the Safety and Efficacy of Fluticasone and Formoterol Combination (FlutiForm™100/10μg and 250/10μg) in a Single Inhaler (SkyePharma HFA MDI) With the Administration of Fluticasone (250μg) and Formoterol (12μg) Concurrently or Alone in Patients With Asthma
Brief Title: Single-dose Crossover Study to Compare the Safety and Efficacy of FlutiForm With Fluticasone and Formoterol Concurrently or Alone in Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Responsible Party: SkyePharma AG, SkyePharma AG
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SKY2028-2-001
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Mild to Moderate Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Formoterol Fumarate; fluticasone-formoterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): * Period 1 Treatment Regimen A: FlutiForm 100/10 ug
  * Period 2 Treatment Regimen B: FlutiForm 250/10 ug
  * Period 3 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug
  * Period 4 Treatment Regimen D: Flixotide Evohaler 250 ug
  Interventions: Drug: fluticasone propionate, formoterol fumarate
- 2 (Active Comparator): * Period 1 Treatment Regimen D: Flixotide Evohaler 250 ug
  * Period 2 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug
  * Period 3 Treatment Regimen B: FlutiForm 250/10 ug
  * Period 4 Treatment Regimen A: FlutiForm 100/10 ug
  Interventions: Drug: fluticasone propionate, formoterol fumarate
- 3 (Active Comparator): * Period 1 Treatment Regimen B: FlutiForm 250/10 ug
  * Period 2 Treatment Regimen A: FlutiForm 100/10 ug
  * Period 3 Treatment Regimen F: Placebo
  * Period 4 Treatment Regimen E: Foradil Aerolizer 12 ug
  Interventions: Drug: fluticasone propionate, formoterol fumarate
- 4 (Active Comparator): * Period 1 Treatment Regimen E: Foradil Aerolizer 12 ug
  * Period 2 Treatment Regimen F: Placebo
  * Period 3 Treatment Regimen A: FlutiForm 100/10 ug
  * Period 4 Treatment Regimen B: FlutiForm 250/10 ug
  Interventions: Drug: fluticasone propionate, formoterol fumarate
- 5 (Active Comparator): * Period 1 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug
  * Period 2 Treatment Regimen D: Flixotide Evohaler 250 ug
  * Period 3 Treatment Regimen E: Foradil Aerolizer 12 ug
  * Period 4 Treatment Regimen F: Placebo
  Interventions: Drug: fluticasone propionate, formoterol fumarate
- 6 (Active Comparator): * Period 1 Treatment Regimen F: Placebo
  * Period 2 Treatment Regimen E: Foradil Aerolizer 12 ug
  * Period 3 Treatment Regimen D: Flixotide Evohaler 250 ug
  * Period 4 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug
  Interventions: Drug: fluticasone propionate, formoterol fumarate

INTERVENTIONS:
Drug: fluticasone propionate, formoterol fumarate — * Period 1 Treatment Regimen E: Foradil Aerolizer 12 ug (One inhalation of formoterol 12 ug)
  * Period 2 Treatment Regimen F: Placebo (Two actuations of Placebo HFA pMDI
  * Period 3 Treatment Regimen A: FlutiForm 100/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 50/5 ug/actuation)
  * Period 4 Treatment Regimen B: FlutiForm 250/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 125/5 ug/actuation)
  Other Names: FlutiForm
  Arms: 1
Drug: fluticasone propionate, formoterol fumarate — * Period 1 Treatment Regimen D: Flixotide Evohaler 250 ug (Two actuations of fluticasone HFA pMDI 125ug/actuation)
  * Period 2 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug (Two actuations of fluticasone HFA pMDI 125ug/actuation and one inhalation of formoterol DPI 12ug/inhalation)
  * Period 3 Treatment Regimen B: FlutiForm 250/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 125/5 ug/actuation)
  * Period 4 Treatment Regimen A: FlutiForm 100/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 50/5 ug/actuation)
  Other Names: FlutiForm
  Arms: 2
Drug: fluticasone propionate, formoterol fumarate — * Period 1 Treatment Regimen B: FlutiForm 250/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 125/5 ug/actuation)
  * Period 2 Treatment Regimen A: FlutiForm 100/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 50/5 ug/actuation)
  * Period 3 Treatment Regimen F: Placebo (Two actuations of placebo HFA pMDI)
  * Period 4 Treatment Regimen E: Foradil Aerolizer 12 ug (One inhalation of formoterol DPI 12 ug)
  Other Names: FlutiForm
  Arms: 3
Drug: fluticasone propionate, formoterol fumarate — * Period 1 Treatment Regimen E: Foradil Aerolizer 12 ug (One inhalation of formoterol DPI 12 ug)
  * Period 2 Treatment Regimen F: Placebo (Two actuations of Placebo HFA pMDI)
  * Period 3 Treatment Regimen A: FlutiForm 100/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 50/5 ug/actuation)
  * Period 4 Treatment Regimen B: FlutiForm 250/10 ug (Two actuations of fluticasone/formoterol HFA pMDI 125/5 ug/actuation)
  Other Names: FlutiForm
  Arms: 4
Drug: fluticasone propionate, formoterol fumarate — * Period 1 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug (Two actuations of fluticasone HFA pMDI 125ug/actuation and one inhalation of formoterol DPI 12ug/inhalation)
  * Period 2 Treatment Regimen D: Flixotide Evohaler 250 ug (Two actuations of fluticasone HFA pMDI 125 ug/actuation)
  * Period 3 Treatment Regimen E: Foradil Aerolizer 12 ug (One inhalation of formoterol DPI 12 ug)
  * Period 4 Treatment Regimen F: Placebo (Two actuations of Placebo HFA pMDI)
  Other Names: FlutiForm
  Arms: 5
Drug: fluticasone propionate, formoterol fumarate — * Period 1 Treatment Regimen F: Placebo (Two actuations of Placebo HFA pMDI
  * Period 2 Treatment Regimen E: Foradil Aerolizer 12 ug (One inhalation of formoterol DPI 12 ug)
  * Period 3 Treatment Regimen D: Flixotide Evohaler 250 ug (Two actuations of fluticasone HFA MDI 125 ug)
  * Period 4 Treatment Regimen C: Flixotide Evohaler 250 ug + Foradil Aerolizer 12 ug (Two actuations of fluticasone HFA pMDI 125ug/actuation and one inhalation of formoterol DPI 12ug/inhalation)
  Other Names: FlutiForm
  Arms: 6

SUMMARY:
The primary purpose was to evaluate the efficacy of SKP FlutiForm HFA MDI compared to placebo or fluticasone and formoterol administered concurrently or alone in asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented history of mild to moderate asthma currently taking a stable dose of inhaled corticosteroid

Exclusion Criteria:

* Smoking history within the last 12 months
* No history of respiratory tract infection within 4 weeks
* No history or evidence of any clinically significant disease or abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-10; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Actual FEV1, % change from Baseline in Actual FEV1, change from Baseline in FEV1 % predicted normal, FEV1 max and FEV1 AUC above the Baseline | pre-dose and at 5, 15, 30, 45, 60, 90 minutes and 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose

SECONDARY OUTCOMES:
Treatment-emergent AEs, clinical laboratory data, 12-lead ECGs and vital signs | 10 weeks including pre- and post-study assessments

CONTACTS AND LOCATIONS:
Overall Officials: SKP, Study Director — SkyePharma AG
Locations (6):
- Investigational site, Belfast, Ireland
- United Kingdom (5):
  - Investigational site, Derbyshire
  - Investigational site, London
  - Investigational site, Manchester
  - Investigational site, Plymouth
  - Investigational site, Slough